CLINICAL TRIAL: NCT01319773
Title: Study of Two Formulations of Cyclosporine Ophthalmic Emulsion in Healthy Volunteers and in Patients With Dry Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 192371-021
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- cyclosporine ophthalmic emulsion Formulation A (Formulation A) (Experimental): Parallel-Group Phase (PGP): cyclosporine ophthalmic emulsion Formulation A
  Interventions: Drug: cyclosporine ophthalmic emulsion Formulation A
- cyclosporine ophthalmic emulsion Formulation B (Formulation B) (Experimental): PGP: cyclosporine ophthalmic emulsion Formulation B
  Interventions: Drug: cyclosporine ophthalmic emulsion Formulation B
- Formulation A and cyclosporine ophthalmic emulsion 0.05% (Other): Paired-Eye Phase (PEP): cyclosporine ophthalmic emulsion Formulation A and cyclosporine ophthalmic emulsion 0.05%
  Interventions: Drug: cyclosporine ophthalmic emulsion Formulation A; cyclosporine ophthalmic emulsion 0.05%
- Formulation B and cyclosporine ophthalmic emulsion 0.05% (Other): PEP: cyclosporine ophthalmic emulsion Formulation B and cyclosporine ophthalmic emulsion 0.05%
  Interventions: Drug: cyclosporine ophthalmic emulsion Formulation B; cyclosporine ophthalmic emulsion 0.05%
- Formulation A and Formulation B (Experimental): PEP: cyclosporine ophthalmic emulsion Formulation A and cyclosporine ophthalmic emulsion Formulation B
  Interventions: Drug: cyclosporine ophthalmic emulsion Formulation A; cyclosporine ophthalmic emulsion Formulation B

INTERVENTIONS:
Drug: cyclosporine ophthalmic emulsion Formulation A — One drop of cyclosporine ophthalmic emulsion Formulation A administered to each eye twice daily for 2 days and once in the morning of Day 3.
  Arms: cyclosporine ophthalmic emulsion Formulation A (Formulation A)
Drug: cyclosporine ophthalmic emulsion Formulation B — One drop of cyclosporine ophthalmic emulsion Formulation B administered to each eye twice daily for 2 days and once in the morning of Day 3.
  Arms: cyclosporine ophthalmic emulsion Formulation B (Formulation B)
Drug: cyclosporine ophthalmic emulsion Formulation A; cyclosporine ophthalmic emulsion 0.05% — One drop of cyclosporine ophthalmic emulsion Formulation A administered to one eye and one drop of cyclosporine ophthalmic emulsion 0.05% administered to the opposite eye, twice daily for 1 day.
  Other Names: RESTASIS®
  Arms: Formulation A and cyclosporine ophthalmic emulsion 0.05%
Drug: cyclosporine ophthalmic emulsion Formulation B; cyclosporine ophthalmic emulsion 0.05% — One drop of cyclosporine ophthalmic emulsion Formulation B administered to one eye and one drop of cyclosporine ophthalmic emulsion 0.05% administered to the opposite eye, twice daily for 1 day.
  Other Names: RESTASIS®
  Arms: Formulation B and cyclosporine ophthalmic emulsion 0.05%
Drug: cyclosporine ophthalmic emulsion Formulation A; cyclosporine ophthalmic emulsion Formulation B — One drop of cyclosporine ophthalmic emulsion Formulation A administered to one eye and one drop of cyclosporine ophthalmic emulsion Formulation B administered to the opposite eye, twice daily for 1 day.
  Arms: Formulation A and Formulation B

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of two formulations of cyclosporine ophthalmic emulsion in healthy adults (parallel-group phase). The parallel-group phase will be followed by a paired-eye phase which will evaluate the safety and tolerability of two formulations of cyclosporine ophthalmic emulsion compared with cyclosporine ophthalmic emulsion (RESTASIS®) in patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

Parallel-Group Phase:

* Weigh at least 110 lbs
* 18 to 45 years old

Paired-Eye Phase:

* Dry eye disease in both eyes

Exclusion Criteria:

Parallel-Group Phase:

* Use of nicotine products, any medications, supplements or herbal products or consumption of grapefruit juice within 14 days or anticipated use during the study
* Has donated blood within 90 days
* Significant weight change (over 10 lbs) within 60 days
* Previous use of RESTASIS®

Parallel-Group and Paired-Eye Phases:

* Anticipated wearing of contact lenses during the study or wearing of contact lenses within 14 days
* Consumption of alcohol products within 72 hours

Paired-Eye Phase:

* Previous ocular surgery
* Use of RESTASIS® within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a parallel-group phase (PGP) and a paired-eye phase (PEP). The paired-eye phase of the study began after the parallel-group phase completed. The parallel-group phase enrolled healthy volunteers and the paired-eye phase enrolled patients with dry eye symptoms.
Groups:
- PGP: Cyclosporine Formulation A: Parallel-Group Phase (PGP): cyclosporine ophthalmic emulsion Formulation A
- PGP: Cyclosporine Formulation B: PGP: cyclosporine ophthalmic emulsion Formulation B
- PEP: Cyclosporine Formulation A and Cyclosporine 0.05%: Paired-Eye Phase (PEP): cyclosporine ophthalmic emulsion Formulation A and cyclosporine ophthalmic emulsion 0.05%
- PEP: Cyclosporine Formulation B and Cyclosporine 0.05%: PEP: cyclosporine ophthalmic emulsion Formulation B and cyclosporine ophthalmic emulsion 0.05%
- PEP: Cyclosporine Formulation A and Cyclosporine Formulation B: PEP: cyclosporine ophthalmic emulsion Formulation A and cyclosporine ophthalmic emulsion Formulation B
Period: Overall Study
Arm/Group | PGP: Cyclosporine Formulation A | PGP: Cyclosporine Formulation B | PEP: Cyclosporine Formulation A and Cyclosporine 0.05% | PEP: Cyclosporine Formulation B and Cyclosporine 0.05% | PEP: Cyclosporine Formulation A and Cyclosporine Formulation B
Started | 10 | 10 | 8 | 8 | 8
Completed | 10 | 10 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PGP: Cyclosporine Formulation A | PGP: Cyclosporine Formulation B | PEP: Cyclosporine Formulation A and Cyclosporine 0.05% | PEP: Cyclosporine Formulation B and Cyclosporine 0.05% | PEP: Cyclosporine Formulation A and Cyclosporine Formulation B | Total
Number analyzed (Participants) | 10 | 10 | 8 | 8 | 8 | 44
Age, Customized [Number; unit: participants]
  18 to 30 years | 8 | 8 | 1 | 1 | 1 | 19
  > 30 to 40 years | 2 | 2 | 0 | 1 | 0 | 5
  > 40 years | 0 | 0 | 7 | 6 | 7 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 5 | 8 | 26
  Male | 7 | 5 | 3 | 3 | 0 | 18

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Cyclosporine Measured in Blood at Day 1 in the Parallel-Group Phase (PGP)
Description: Concentration of cyclosporine measured in blood at Day 1 of the parallel-group phase (PGP). Blood samples were collected up to 3 hours post-dose and concentrations of cyclosporine were measured.
Time Frame: Day 1
Population: Safety Population: All randomized subjects who were treated with at least 1 dose of study medication.
Measure: Number; unit: Nanogram/milliliter (ng/mL)
Arm/Group | Cyclosporine Formulation A | Cyclosporine Formulation B
Number analyzed (Participants) | 10 | 10
Nanogram/milliliter (ng/mL)
  Time = pre-dose | NA — Below limit of quantification | NA — Below limit of quantification
  Time = 0.5 hours | NA — Below limit of quantification | NA — Below limit of quantification
  Time = 1 hour | NA — Below limit of quantification | NA — Below limit of quantification
  Time = 3 hours | NA — Below limit of quantification | NA — Below limit of quantification

2. Secondary Outcome: Number of Subjects Who Reported Ocular Symptoms During the Parallel-Group Phase (PGP)
Description: Number of subjects who reported ocular symptoms of any severity during the parallel-group phase (PGP) of the study. Subjects evaluated the presence and severity of ocular symptoms in each eye. The severity of each symptom (blurring, foreign body sensation, pain, burning/stinging, tearing, and itching) were recorded on a 5-point scale (0=none, +0.5=very mild,+1=mild, +2=moderate, and +3=severe).
Time Frame: 3 Days
Population: Per Protocol: All randomized subjects who received their assigned study medication and closely followed the protocol.
Measure: Number; unit: Number of Subjects
Arm/Group | Cyclosporine Formulation A | Cyclosporine Formulation B
Number analyzed (Participants) | 10 | 10
Number of Subjects | 3 | 1

3. Secondary Outcome: Number of Eyes With Ocular Symptoms Post-Dose During the Paired-Eye Phase (PEP) at Day 1
Description: Number of eyes with ocular symptoms of any severity, post-dose in the paired-eye phase (PEP) at Day 1. Subjects evaluated the presence and severity of ocular symptoms in each eye. The severity of each symptom (blurring, foreign body sensation, pain, burning/stinging, tearing, and itching) were recorded on a 5-point scale (0=none, +0.5=very mild, +1=mild, +2=moderate, and +3=severe).
Time Frame: Day 1
Population: Per Protocol: All randomized subjects who received their assigned study medication and closely followed the protocol.
Measure: Number; unit: Number of Eyes
Units Other Than Participants: Eyes
Arm/Group | Cyclosporine Formulation A | Cyclosporine Formulation B | Cyclosporine 0.05%
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (Eyes) | 16 | 16 | 16
Number of Eyes
  Blurring | 2 | 1 | 1
  Foreign Body Sensation | 0 | 0 | 0
  Pain | 0 | 1 | 0
  Burning/Stinging | 3 | 2 | 2
  Tearing | 1 | 2 | 3
  Itching | 0 | 0 | 0

ADVERSE EVENTS:
Description: SAEs and AEs are reported by treatment assignment or arm as randomized not by individual intervention received.
Arm/Group | PGP: Cyclosporine Formulation A | PGP: Cyclosporine Formulation B | PEP: Cyclosporine Formulation A and Cyclosporine 0.05% | PEP: Cyclosporine Formulation B and Cyclosporine 0.05% | PEP: Cyclosporine Formulation A and Cyclosporine Formulation B
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10 | 5/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PGP: Cyclosporine Formulation A (N=10) | PGP: Cyclosporine Formulation B (N=10) | PEP: Cyclosporine Formulation A and Cyclosporine 0.05% (N=8) | PEP: Cyclosporine Formulation B and Cyclosporine 0.05% (N=8) | PEP: Cyclosporine Formulation A and Cyclosporine Formulation B (N=8)
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Punctate Keratitis (Eye disorders) | 1 | 2 | 2 | 1 | 0
Conjunctival Hyperaemia (Eye disorders) | 1 | 0 | 4 | 4 | 6
Abnormal Sensation in Eye (Eye disorders) | 0 | 0 | 1 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eyelid Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 5 | 2
Eye Pain (Eye disorders) | 0 | 0 | 0 | 3 | 1
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 2 | 3
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 2 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 2
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 1 | 1
Dysguesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo